CLINICAL TRIAL: NCT05865600
Title: Perfusion Estimation for Optimal Revascularization and Medical Therapy in Chronic Coronary Syndrome - a Randomized Trial
Brief Title: Perfusion Estimation For Optimal Treatment Strategy in Chronic Coronary Syndrome
Acronym: PERFORM-CCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Gødstrup Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-10-72-185-22
Record Dates: First submitted 2023-05-02; First posted 2023-05-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-08

CONDITIONS: Chronic Coronary Syndrome; Myocardial Ischemia; Stable Angina; Coronary Artery Disease
Keywords: Myocardial Ischemia; Angina Pectoris; Coronary Artery Disease; Coronary Angiography; Computed Tomography Angiography; Myocardial Perfusion Imaging
MeSH Terms: conditions — Myocardial Ischemia; Angina, Stable; Coronary Artery Disease; Angina Pectoris | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: All eligible patients are included in a prospective cohort with repeated questionnaires.
  Patients with abnormal perfusion and clinical indication for invasive coronary angiography are randomized 1:1 in permuted blocks with random varying sizes of 4,6 and 8 to either immediate invasive coronary angiography or delayed invasive coronary angiography via a standard computerized random-number generator stratified for age ≥70 years and sex (REDcap). Proper concealment of randomization is obtained by the use of an external randomization service (Clinical Trial Unit, Dept. of Clinical Medicine, Aarhus University, Denmark).
Masking Description: Patients will be blinded to the specific result of the initial [15O]H2O cardiac PET/CT. The result will be reported as normal, abnormal, or suspicion of unprotected left main coronary stenosis (exclusion criteria) until the termination of the study. Investigators and invasive coronary angiography operators are not blinded to the specific result of the initial [15O]H2O cardiac PET/CT in order to evaluate clinical indication for invasive coronary angiography. The coronary CT angiography will only be evaluated for unprotected left main coronary artery stenosis - the rest of the coronary CT angiography as well as the two additional [15O]H2O cardiac PET/CT scans at 3 and 6 months assessment will only be analyzed after the termination of the study. Investigators will be blinded to the results of baseline, 3, and 6 month questionnaires and walking distances until the termination of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort study (Other): All patients with symptomatic chronic coronary syndrome undergoing clinically referred [15O]H2O cardiac PET/CT will be included in a prospective cohort with repeated symptom questionnaires and outcomes registered in national registries. A total of 570 patients are expected to be included in order to have 200 randomized patients reaching the 3-month assessment
  Interventions: Other: Standard of care
- Immediate referral to invasive coronary angiography (Experimental): Patients with abnormal perfusion on [15O]H2O cardiac PET/CT and clinical indication for invasive coronary angiography randomized to immediate referral for invasive coronary angiography with concomitant optimization of guideline-directed medical therapy. Enrollment will continue until a total of 200 randomized patients reach the 3-month assessment.
  Interventions: Other: Optimization of guideline-directed medical therapy; Diagnostic Test: Immediate referral for invasive coronary angiography
- Delayed referral to invasive coronary angiography (Experimental): Patients with abnormal perfusion on [15O]H2O cardiac PET/CT and clinical indication for invasive coronary angiography randomized to 3-months delayed referral for invasive coronary angiography with concomitant optimization of guideline-directed medical therapy. Enrollment will continue until a total of 200 randomized patients reach the 3-month assessment.
  Interventions: Other: Optimization of guideline-directed medical therapy; Diagnostic Test: 3-months delayed referral for invasive coronary angiography

INTERVENTIONS:
Other: Optimization of guideline-directed medical therapy — Consultation every second week with optimization of guideline-directed medical therapy according to 2019 ESC guidelines on chronic coronary syndrome. Focus will be on risk-factor modification and anti-anginal medication with the treatment aim to achieve freedom from angina and dyspnea with a heart rate at rest ≤ 60 beats/min and systolic blood pressure > 100 mmHg.
  Arms: Delayed referral to invasive coronary angiography; Immediate referral to invasive coronary angiography
Diagnostic Test: Immediate referral for invasive coronary angiography — Immediate referral for invasive coronary angiography
  Arms: Immediate referral to invasive coronary angiography
Diagnostic Test: 3-months delayed referral for invasive coronary angiography — 3-months delayed referral for invasive coronary angiography
  Arms: Delayed referral to invasive coronary angiography
Other: Standard of care — Standard of care
  Arms: Cohort study

SUMMARY:
We will establish a cohort of 570 symptomatic chronic coronary syndrome patients undergoing 15O-water PET and assess their symptoms through repeated questionnaires. Two hundred patients with abnormal perfusion will be randomized to immediate or delayed referral to invasive coronary angiography with concomitant optimization of guideline-directed medical therapy with repeated 15O-water PET and questionnaires at 3 and 6 months. The primary objective is to compare the potential benefit of early invasive coronary angiography (ICA) versus guideline directed medical therapy (GDMT) on symptomatic relief defined as freedom of angina after 3 months following a positive [15O]H2O cardiac PET/CT in patients with symptomatic chronic coronary syndrome.

DETAILED DESCRIPTION:
BACKGROUND:

Ischemic heart disease (IHD) is highly prevalent in Western countries and an emerging disease in developing countries around the globe. While the Danish incidence rate of IHD for both females and males has been declining during the last 15 years, the prevalence has stabilized at 165,000 patients in 2018 due to enhanced survival.

Ischemic heart disease is caused by atherosclerotic plaque formation in the epicardial coronary arteries, abnormalities in the coronary microcirculation, spasms in the vessel wall, or a combination thereof. This may result in chest discomfort or dyspnoea leading to frequent primary care consultations and admissions on the suspicion of acute coronary syndrome. To emphasize the chronic nature of the disease, the European Society of Cardiology has replaced the previous nomenclature of stable coronary artery disease with chronic coronary syndrome (CCS) in their latest guidelines from 2019.

When cardiac imaging is used to diagnose and select treatment in patients with CCS, guidelines recommend non-invasive functional imaging modalities in patients with an intermediate or high clinical likelihood of IHD or in patients with prior revascularization. In patients with prior myocardial infarction or percutaneous coronary intervention, studies have found higher diagnostic accuracy of [15O]H2O cardiac PET/CT with measurement of absolute quantification of myocardial perfusion to diagnose obstructive coronary artery disease compared with single-photon emission computed tomography and magnetic resonance imaging. Current European guidelines recommend myocardial revascularization in addition to guideline-directed medical therapy (GDMT) in CCS patients with large areas of ischemia (≥ 10%) in the left ventricle to improve prognosis.

Since the publication of these guidelines, a large randomized trial of initial invasive versus conservative strategy in patients with moderate-severe ischemia on stress testing has been published with no observed prognostic benefit of an initial invasive strategy in these patients. However, patients assigned to an initial invasive strategy had a greater improvement in angina-related health status as compared with a conservative strategy, with larger differences observed in patients who were more symptomatic at baseline. The study is limited by the high use of stress ECG (25% of participants) which has a very low diagnostic power and the high proportion of asymptomatic participants at baseline (35%).

It is unknown whether the results of MPI with absolute quantification of myocardial perfusion can improve the selection of patients with an additional symptomatic benefit of an initial invasive strategy compared with GDMT.

METHODS:

Patients with symptomatic CCS referred for clinically indicated [15O]H2O cardiac PET/CT will be included in a prospective cohort and assessed with questionnaires at baseline, 3, 6, 12, 60, and 120 months. Clinical outcomes will be assessed through national registries.

Patients with abnormal perfusion and a clinical indication for ICA will undergo coronary CT angiography and a six-minute walking test. Hereafter, they will be randomized 1:1 to immediate referral to ICA or 3 months delayed referral to ICA. Both groups will undergo optimization of GDMT with consultations every two weeks.

At 3 and 6 months, both groups will undergo repeated questionnaires, [15O]H2O cardiac PET/CT and a six-minute walking test.

Enrollment in the cohort study and randomized trial will continue until 200 randomized patients have reached the 3 months assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Willing to participate and able to understand, read and sign the informed consent document before the planned procedure
3. Known ischemic heart disease defined as one of the following

   1. Previous myocardial infarction, percutaneous coronary intervention or coronary artery bypass grafting
   2. Previous coronary computed tomography angiography or invasive coronary angiography documenting atherosclerosis.
4. Undergoing clinically indicated [15O]H2O cardiac PET/CT due to chest discomfort or dyspnea as angina equivalent

   Additional inclusion criteria for randomized trial:
5. Initial [15O]H2O cardiac PET/CT with abnormal perfusion defined as all of the following

   1. Hyperemic myocardial blood flow (hMBF) ≤2.3 mL/min/g in at least two adjacent myocardial segments
   2. Relative hMBF ≤ 65% in at least two adjacent segments as compared with the mean hMBF of the two adjacent segments with the highest mean hMBF
   3. Tissue perfusion defect extent ≥ 5% based on indices of relative hypoperfusion
6. Clinical indication for invasive coronary angiography decided at a multidisciplinary conference between consultants in nuclear medicine and cardiology

Exclusion Criteria:

1. Ongoing acute coronary syndrome or acute coronary syndrome within 30 days
2. Contraindications for adenosine

   1. Severe asthma
   2. Advanced atrioventricular block without pacemaker
   3. Severe aortic stenosis
3. Patients not able to breath hold (severe COPD/asthma)
4. Pregnant women, including women who are potentially pregnant or lactating
5. Allergy to iomeron
6. Life expectancy of less than 2 years
7. Severe valvular disease
8. Reduced kidney function with an estimated glomerular filtrations rate <40 ml/min
9. Inability to consent

   Additional exclusion criteria for randomized trial:
10. Unprotected left main coronary artery stenosis on coronary CT angiography
11. Very large perfusion defect on initial [15O]H2O cardiac PET/CT indicating left main coronary artery stenosis or balanced ischemia defined as tissue perfusion defect extent based on indices of absolute hMBF ≥ 20% in two or more myocardial territories supplied by coronary arteries with an Agatston calcium score ≥ 300

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 570 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2026-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Symptomatic relief | After 3 months following a positive [15O]H2O cardiac PET/CT
  Seattle Angina Questionnaire-7 angina frequency score = 100 (0-100 with higher scores indicating less frequent angina)

SECONDARY OUTCOMES:
Walking capacity | 3 and 6 months after randomization
  Meters walked in six-minute walking test
Angina frequency | 3, 6, 12, 60, and 120 months after randomization or index [15O]H2O cardiac PET/CT
  Seattle Angina Questionnaire-7 angina frequency score (0-100 with higher scores indicating less frequent angina)
Physical limitation | 3, 6, 12, 60, and 120 months after randomization or index [15O]H2O cardiac PET/CT
  Seattle Angina Questionnaire-7 physical limitation score (0-100 with higher scores indicating less physical limitation)
Quality of life-score | 3, 6, 12, 60, and 120 months after randomization or index [15O]H2O cardiac PET/CT
  Seattle Angina Questionnaire-7 quality of life score (0-100 with higher scores indicating better quality of life)
Health status | 3, 6, 12, 60, and 120 months after randomization or index [15O]H2O cardiac PET/CT
  Seattle Angina Questionnaire-7 summary score (0-100 where 0 denotes the lowest reportable health status and 100 the highest)
Dyspnea | 3, 6, 12, 60, and 120 months after randomization or index [15O]H2O cardiac PET/CT
  Rose Dyspnea Scale. Scores range from 0 to 4, where 0 indicates no dyspnea with activity and 4 indicates significant limitations due to dyspnea
Work Ischemic Symptom score | 3, 6, 12, 60, and 120 months after randomization or index [15O]H2O cardiac PET/CT
  Work Ischemic Symptom score summary score. The scoring system is currently under development.
Hyperemic myocardial blood flow | 3 and 6 months after randomization
  Global and territorial hyperemic myocardial blood flow (ml/g/min) of perfusable myocardium on [15O]H2O cardiac PET/CT.
Myocardial flow reserve | 3 and 6 months after randomization
  Global and territorial myocardial flow reserve (unitless measure) on [15O]H2O cardiac PET/CT.
Coronary flow capacity | 3 and 6 months after randomization
  Coronary flow capacity incorporates hyperemic myocardial blood flow and myocardial flow reserve into a 5-point ordinal scale ranging from myocardial steal indicating very poor coronary flow capacity to normal coronary flow capacity. All data is derived from [15O]H2O cardiac PET/CT.
Coronary revascularization | 3 and 6 months after randomization or index [15O]H2O cardiac PET/CT
  Percutaneous coronary intervention and/or coronary artery bypass grafting
Coronary revascularization | 10 years after randomization or index [15O]H2O cardiac PET/CT
  Percutaneous coronary intervention and/or coronary artery bypass grafting
Myocardial infarction | 3 and 6 months after randomization or index [15O]H2O cardiac PET/CT
  All myocardial infarctions
Myocardial infarction | 10 years after randomization or index [15O]H2O cardiac PET/CT
  All myocardial infarctions
All-cause mortality | 3 and 6 months after randomization or index [15O]H2O cardiac PET/CT
  All deaths
All-cause mortality | 10 years after randomization or index [15O]H2O cardiac PET/CT
  All deaths
Cardiovascular mortality | 3 and 6 months after randomization or index [15O]H2O cardiac PET/CT
  All cardiovascular deaths
Cardiovascular mortality | 10 years after randomization or index [15O]H2O cardiac PET/CT
  All cardiovascular deaths
Unstable angina | 3 and 6 months after randomization or index [15O]H2O cardiac PET/CT
  Unstable angina
Unstable angina | 10 years after randomization or index [15O]H2O cardiac PET/CT
  Unstable angina
Unplanned hospitalization | 3 and 6 months after randomization or index [15O]H2O cardiac PET/CT
  Any hospitalization requiring overnight stay not electively planned
Unplanned hospitalization | 10 years after randomization or index [15O]H2O cardiac PET/CT
  Any hospitalization requiring overnight stay not electively planned
De novo heart failure | 3 and 6 months after randomization or index [15O]H2O cardiac PET/CT
  New diagnosis of heart failure
De novo heart failure | 10 years after randomization or index [15O]H2O cardiac PET/CT
  New diagnosis of heart failure
Use of CCTA, MPI, and ICA | 10 years after randomization or index [15O]H2O cardiac PET/CT
  Use of coronary CT angiography, myocardial perfusion imaging and invasive coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Morten Böttcher, Prof, Principal Investigator — University Clinic for Cardiovascular Research, Dept. of Cardiology, Gødstrup Hospital
Locations (1):
- Gødstrup Hospital, Herning, Central Jutland, Denmark

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be readily available due to Danish legislation. Data can be shared upon reasonable request if a research protocol is submitted to the investigators and approval for data sharing is obtained via Danish authorities.